CLINICAL TRIAL: NCT01589302
Title: A Phase 2 Study of the Bruton's Tyrosine Kinase (Btk) Inhibitor, PCI-32765(Ibrutinib), in Relapsed and Refractory Patients With Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL) and B-cell Prolymphocytic Leukemia (B-PLL)
Brief Title: PCI-32765 (Ibrutinib) in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia, Small Lymphocytic Lymphoma, or B-cell Prolymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kami Maddocks, MD (Other)
Responsible Party: Sponsor-Investigator, Kami Maddocks, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-11133; NCI-2012-00560 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-04-23; First posted 2012-05-01 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Prolymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory/Relapsed Chronic Lymphocytic Leukemia
Keywords: Bruton's Tyrosine Kinase; CLL; SLL; B-PLL
MeSH Terms: conditions — Leukemia, Prolymphocytic; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib) (Experimental): Patients will be treated with PCI-32765 capsules administered orally once daily at a dose of 420 mg for 28 day cycles. Weekly monitoring during the first month will occur followed by monthly evaluations for 2 additional months. Monitoring for patients at this point would be every 3 months with monthly CBC(complete blood count)and phone follow-up with a co-investigator on the study. A standard questionnaire will be used in this monthly phone assessment. Patients will continue to receive the study drug indefinitely as long as they are deriving clinical benefit (Complete Response or Partial Response or Stable Disease) and not experiencing any unacceptable toxicity. Subjects with disease progression will be removed from the study. Correlative laboratory samples, quality of life assessment, and immunologic data would be collected over time of therapy.
  Interventions: Drug: ibrutinib; Other: Correlative laboratory samples; Other: quality of life assessment

INTERVENTIONS:
Drug: ibrutinib — Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Other Names: Bruton's tyrosine kinase inhibitor PCI-32765; BTK inhibitor PCI-32765; PCI-32765
Other: Correlative laboratory samples — Blood samples will be collected and used for pharmacodynamic testing. Samples will be collected pre-dose on Cycle 1 Day 1 and 2 hours post-dose Cycle 1 Day 1, pre-dose on Day 2 and Day 8 of Cycle 1 and pre-dose on Day 1 of Cycles 2 and 3 and then every 3 cycles thereafter for 1 year (Cycle 15 Day 1). Samples will also be collected at the time of relapse and at any time when bone marrow biopsy is performed.
  Other Names: laboratory biomarker anyalysis
Other: quality of life assessment — During screening, sociodemographic information (e.g., age, race, marital status) and reports of recent (last year) stressful events will be obtained. The assessment will consist of measures of emotional distress, depressive symptoms, and quality of life. Quality of life measures will be administered during screening and on Days 1 (±3), 8 (±3),, 15 (±3),, 22 (±3), of Cycle 1, Day 1 (±3), of Cycle 2 and on day 1 (±7) of Cycles 3, 6, and then every 3 months thru month 24.

SUMMARY:
This is a Phase II, single institution open-label, non-randomized monotherapy study to evaluate the clinical efficacy and durable disease control of PCI-32765 administered to patients with relapsed/refractory CLL/SLL/PLL of all risk categories with patients having deletion 17p13 independently evaluated.

DETAILED DESCRIPTION:
This is a clinical trial, a type of research study, involving treatment with an investigational (experimental) drug called PCI-32765 (Ibrutinib), a "kinase inhibitor". "Kinases" are proteins that are inside of cells and help them to live and grow. The specific kinase inhibited or blocked by this study drug is believed to help blood cancer cells grow and live. By inhibiting or "blocking" the activity of this kinase, it is possible that the study drug may be able to kill the cancer cells or stop them from growing. This study will involve treating patients with chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), or B-cell prolymphocytic leukemia (B-PLL) that has not responded to or has relapsed after standard treatment. This trial is studying how effective PCI-32765 is at treating CLL, SLL, or B-PLL and all the effects, good and/or bad, treatment with this drug has on patients and their cancers.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of relapsed/refractory CLL/SLL who require treatment and have failed at least one prior therapy.
* Patients must have available results of interphase cytogenetics CLL fluorescent in situ hybridization (FISH) panel; the cytogenetic analysis must be done prior to starting therapy but after any recent therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy greater than 2 months
* Bilirubin =< 1.5 X the institutional upper limit of normal unless due to Gilbert's disease or disease related to Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 X the institutional upper limit of normal unless disease related
* Creatinine =< 1.5 X the institutional upper limit of normal unless disease related
* Absolute neutrophil count (ANC) >= 0.75 X 10^9/L
* Platelet count >= 30 X 10^9/L
* Agree to use contraception during the study and for 30 days after the last dose of study drug if sexually active and able to bear children
* Ability to understand and the willingness to sign a written informed consent document
* Patients with uncontrolled or active infection requiring antibiotic therapy; patients with controlled infections who are receiving extended antibiotics or prophylactic therapy are not excluded

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy or immunotherapy within 4 weeks prior to the first dose of study drug (corticosteroids for disease-related symptoms allowed but doses equivalent to > 20 mg prednisone orally per day require 1 week washout before study drug administration or steroid dose must be equal to =< 20 mg prednisone orally daily)
* Patients who have not recovered from adverse events of >= grade 3 toxicity due to agents administered more than 4 weeks ago
* Receiving any other investigational agents
* Previously randomized to any PCI-32765 clinical trial
* Known secondary malignancy that limits survival to less than two years
* Patients with malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
* Patients requiring anti-coagulation with warfarin or other Vitamin K antagonists or heparin products including low molecular weight heparin (LMWH)
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification
* Patients requiring treatment with a strong cytochrome P450 3A4/5 (CYP3A4/5) and/or cytochrome P450 2D6 (CYP2D6) inhibitor
* Patients with a life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of PCI-32765 PO, or put the study outcomes at undue risk
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Active central nervous system (CNS) involvement by lymphoma
* Pregnant or women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-05-21 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kami Maddocks, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Arrato NA, Valentine TR, Byrd JC, Jones JA, Maddocks KJ, Woyach JA, Andersen BL. Illness representations and psychological outcomes in chronic lymphocytic leukaemia. Br J Health Psychol. 2022 May;27(2):553-570. doi: 10.1111/bjhp.12562. Epub 2021 Oct 4. PMID 34608724
- [Derived] Long M, Beckwith K, Do P, Mundy BL, Gordon A, Lehman AM, Maddocks KJ, Cheney C, Jones JA, Flynn JM, Andritsos LA, Awan F, Fraietta JA, June CH, Maus MV, Woyach JA, Caligiuri MA, Johnson AJ, Muthusamy N, Byrd JC. Ibrutinib treatment improves T cell number and function in CLL patients. J Clin Invest. 2017 Aug 1;127(8):3052-3064. doi: 10.1172/JCI89756. Epub 2017 Jul 17. PMID 28714866
- [Derived] Maddocks KJ, Ruppert AS, Lozanski G, Heerema NA, Zhao W, Abruzzo L, Lozanski A, Davis M, Gordon A, Smith LL, Mantel R, Jones JA, Flynn JM, Jaglowski SM, Andritsos LA, Awan F, Blum KA, Grever MR, Johnson AJ, Byrd JC, Woyach JA. Etiology of Ibrutinib Therapy Discontinuation and Outcomes in Patients With Chronic Lymphocytic Leukemia. JAMA Oncol. 2015 Apr;1(1):80-7. doi: 10.1001/jamaoncol.2014.218. PMID 26182309
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Ibrutinib): Patients were treated with PCI-32765 capsules administered orally once daily at a dose of 420 mg for 28 day cycles. Patients will continue to receive the study drug indefinitely as long as they are deriving clinical benefit and not experiencing any unacceptable toxicity. Subjects with disease progression will be removed from the study. Correlative laboratory samples, quality of life assessment, and immunologic data would be collected over time of therapy. Patients received ibrutinib orally (PO) once daily(QD)on days 1-28. Courses repeat every 28 days in the absence of disease progression
Period: Overall Study
Arm/Group | Treatment (Ibrutinib)
Started (2 patients were not eligible for study and did not being treatment) | 154
Del17p Patients | 76
Non-Del17p Patients | 76
Completed | 152
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 152
Age, Continuous [Median (Full Range); unit: years]
  Del17p patients | 66 [42 to 91]
  Non-Del17p patients | 64 [26 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 108
Region of Enrollment [Number; unit: patients]
  United States | 152

OUTCOME MEASURES:

1. Primary Outcome: Determine the 2 Year Progression-free Survival (PFS) of Single Agent PCI-32765 in Patients With Relapsed and Refractory CLL.
Description: We will summarize our findings for this endpoint independently as well within each cohort (del17p vs other cytogenetic groups). We will evaluate the proportion of patients who are progression-free and alive at two years or have gone on to transplant (treatment successes) over the total number of evaluable patients; eligible patients who received at least one dose of therapy are considered evaluable. Assuming that the number of treatment successes as defined above is binomially distributed, we will also include 95% binomial confidence intervals for the estimates corresponding to each cohort.
Time Frame: up to 2 years
Population: There are 2 different cohorts Del (17p) and Non-Del (17p) each with 76 patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Treatment (Ibrutinib): Patients treated with PCI-32765 capsules administered orally once daily at a dose of 420 mg for 28 day cycles. Weekly monitoring during the first month will occur followed by monthly evaluations for 2 additional months. Monitoring for patients at this point would be every 3 months with monthly CBC(complete blood count)and phone follow-up with a co-investigator on the study. A standard questionnaire will be used in this monthly phone assessment. Patients will continue to receive the study drug indefinitely as long as they are deriving clinical benefit (Complete Response or Partial Response or Stable Disease) and not experiencing any unacceptable toxicity. Subjects with disease progression will be removed from the study. Correlative laboratory samples, quality of life assessment, and immunologic data would be collected over time of therapy.
  ibrutinib: Patients received ibrutinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 152
percentage of patients
  All patients | 64 [57 to 72]
  Del(17p): number analyzed (Participants) | 76
  Del(17p) | 64 [54 to 75]
  non-Del(17p): number analyzed (Participants) | 76
  non-Del(17p) | 64 [54 to 75]

2. Secondary Outcome: Best Overall Response Rate Using the Revised International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Working Group Guidelines
Description: Responders were subjects who achieved a complete response (CR), partial response (PR) or PR with persistent lymphocytosis. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: up to 2 years
Population: There are 2 different cohorts Del (17p) and Non-Del (17p) each with 76 patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 152
percentage of patients
  All patients | 63 [55 to 70]
  Del(17p): number analyzed (Participants) | 76
  Del(17p) | 66 [55 to 76]
  non-Del(17p): number analyzed (Participants) | 76
  non-Del(17p) | 59 [48 to 70]

3. Secondary Outcome: Number of Patients With 6 Month ORR of Single Agent Ibrutinib in Relapsed and Refractory CLL Patients
Description: The 6 month overall response rates overall response rate (ORR). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 6 months
Population: There are 2 different cohorts Del (17p) and Non-Del (17p) each with 76 patients
Measure: Number (95% Confidence Interval); unit: patients
Groups:
- Treatment (Ibrutinib): Patients will be treated with PCI-32765 capsules administered orally once daily at a dose of 420 mg for 28 day cycles. Weekly monitoring during the first month will occur followed by monthly evaluations for 2 additional months. Monitoring for patients at this point would be every 3 months with monthly CBC(complete blood count)and phone follow-up with a co-investigator on the study. A standard questionnaire will be used in this monthly phone assessment. Patients will continue to receive the study drug indefinitely as long as they are deriving clinical benefit (Complete Response or Partial Response or Stable Disease) and not experiencing any unacceptable toxicity. Subjects with disease progression will be removed from the study. Correlative laboratory samples, quality of life assessment, and immunologic data would be collected over time of therapy.
  ibrutinib: Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease pro
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 152
patients
  All patients | 63 [55 to 70]
  Del(17p): number analyzed (Participants) | 76
  Del(17p) | 66 [55 to 76]
  Non-del(17p): number analyzed (Participants) | 76
  Non-del(17p) | 59 [48 to 70]

4. Secondary Outcome: Percentage of Patients With Overall Survival (OS)
Description: Time from date of first treatment with ibrutinib until the date of death from any cause or the date of last contact for those alive.
Time Frame: 2 years
Population: There are 2 different cohorts Del (17p) and Non-Del (17p) each with 76 patients
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 152
percent of patients
  All patients | 78 [71 to 84]
  Del(17p): number analyzed (Participants) | 76
  Del(17p) | 75 [63 to 83]
  non-Del(17p): number analyzed (Participants) | 76
  non-Del(17p) | 81 [71 to 89]

5. Secondary Outcome: 2-year Kaplan-Meier Estimate of OS for Relapsed and Refractory CLL Patients Treated With Single Agent PCI-32765
Description: Time from date of first treatment with ibrutinib until the date of progression or death from any cause. Those alive and progression free are censored at the date of last clinical assessment.
Time Frame: 2 years
Population: There are 2 different cohorts Del (17p) and Non-Del (17p) each with 76 patients
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 152
percent of patients
  All patients | 69 [61 to 76]
  Del(17p): number analyzed (Participants) | 76
  Del(17p) | 66 [54 to 76]
  non-Del(17p): number analyzed (Participants) | 76
  non-Del(17p) | 72 [60 to 81]

6. Secondary Outcome: Number of Patients With Adverse Events, Graded According to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Adverse events grade 3 or higher using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 with the attribution of either definite, possible or probable related.
Time Frame: Up to 2 years post treatment
Measure: Number; unit: patients
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 152
patients
  Anemia | 13
  Febrible Neutropenia | 2
  Leukocytosis | 18
  Atrial Fibrillation | 1
  Diarrhea | 2
  Gastric Hemorrhage | 1
  Gastrointestinal Disorders-other | 1
  Mucositis Oral | 1
  Nausea | 2
  Death | 1
  Edema Limb | 1
  Fatigue | 1
  General Disorders and Admin Site Conditions | 2
  Cholecystitis | 1
  Bronchial Infection | 1
  Infections and Infestations-other | 4
  Lung Infection | 10
  Otitis Media | 1
  Sepsis | 2
  Skin Infection | 2
  Urinary Tract Infection | 1
  Alanine Aminotransferase Increased | 1
  Blood Bilirubin Increased | 1
  Lymphocyte Count Decreased | 14
  Lymphocyte Count Increased | 54
  Neutrophil Count Decreased | 40
  Platelet Count Decreased | 8
  White Blood Cell Decreased | 10
  Hyperuricemia | 4
  Hypophosphatemia | 1
  Arthralgia | 2
  Arthritis | 1
  Hematuria | 2
  Hypoxia | 1
  Respiratory Failure | 1
  Rash Maculo-papular | 1
  Hematoma | 1
  Hypertension | 7

7. Secondary Outcome: Resistance Studies of Ibrutinib
Description: Percentage of patients with BTK C481S mutation or PLCG2 mutation
Time Frame: Up to 4 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 152
percentage of patients | 13.2 [8.2 to 19.6]

8. Secondary Outcome: Decrease in Immune Suppression of CLL Cells
Time Frame: up to 3 months
Population: Data was not collect and analyzed for this outcome measure
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 0

9. Secondary Outcome: Effectiveness of Ibrutinib Bridging Patients to Allogeneic Stem Cell Transplant and Outcome of Patients Following This Intervention
Description: The number of participants with successful Allogenic Stem Cell Transplant
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 152
participants | 1

10. Secondary Outcome: Cancer-Specific Stress as Measured by the Impact of Event Scale-Revised (IES-R)
Description: Cancer-Specific Stress was measured by the Impact of Event Scale-Revised Participants rated the intensity of these feelings using a five-point Likert scale ranging from 0=not at all to 4=extremely. Patients rated the frequency of their feelings or events for the previous week before treatment. The items were summed for a total score that ranged from 0 to 64
Time Frame: Up to 2 years
Population: Data was reported for start of treatment only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 152
units on a scale | 9.18 (8.35)

11. Secondary Outcome: Cognitive-Affective Depressive Symptoms as Measured by the Beck Depression Inventory-2nd Edition (BDI-II)
Description: The Beck Depression Inventory-2nd edition is a 21-item measure of depressive symptoms. Scores were calculated representing the cognitive-affective and the somatic symptoms associated with depression (e.g. sadness, pessimism, loss of pleasure) during past month on scale from 0 to 3. Items were summed, with higher scores indicating more depressive symptoms. The scores on the scale from range from 0 to 42.
Time Frame: at 5 months
Population: Data was reported for month 5 from start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 130
units on a scale | 1.88 (3.11)

12. Secondary Outcome: Negative Mood Quality of Life Measured by a 37-item Questionnaire
Description: The Profile of Mood States-Short Form (POMS-SF) yields six subscales, Tension, Depression, Anger, Vigor, Fatigue, and Confusion. A total mood disturbance score is found by summing the six subscales. Total Mood Disturbance (TMD) scores range from -24 to 124 with higher scores indicating greater mood disturbance.
Time Frame: at 5 months
Population: Data was reported for month 5 from start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 128
units on a scale | 0.89 (18.12)

13. Secondary Outcome: Mental Health Quality of Life Was Measured by the Mental Component Summary Score of the Medical Outcomes Study
Description: SF-12 assesses aspects of quality of life including physical functioning, role functioning-physical, bodily pain, general health perceptions, vitality, social functioning, role functioning-emotional, and mental health. Subscale raw scores are transformed to put each subscale on a 0-100 range with higher scores indicative of greater functioning. Subscale scores are standardized based on US General Population norms and aggregated based on factor score coefficients into two component scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Component scores are norm-based t-scores meaning scores above 50 indicate better functioning than average functioning while scores below 50 indicate worse functioning.
Time Frame: at 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 126
units on a scale | 53.98 (8.72)

14. Secondary Outcome: Fatigue Symptom Inventory (FSI) Interference Quality of Life as Measured by a 11-item Total Disruption Index Sub Scale of Fatigue Symptoms Inventory
Description: The Fatigue Interference quality of life measures is a 11-item self reported questionnaire used to measure frequency, severity and daily pattern of fatigue Symptoms as well as impact of QOL in the past week. The Total Disruption Index (TDI) an 7 item subset of FSI was used. Items were rated on a 11-point Likert scale from 0=no interference to 10=extreme interference. Total scores could range from 0 to 70, with higher scores indicating greater fatigue interference.
Time Frame: at 5 months
Population: Data was reported for month 5 from the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 129
units on a scale | 9.70 (13.11)

15. Secondary Outcome: Sleep Through Quality of Life as Measured by a Medical Outcomes Study-Sleep Scale
Description: Sleep problems quality of life measures is a six-item sleep problems index I of the Medical Outcomes Study-Sleep Scale used to assess sleep problems. Participants reported how often they experience six specific difficulties with sleep on a 6-point Likert scale (1=All of the time to 6=None of the time). Scores transformed into a 0-100 scale with higher scores indicating greater sleep problems.
Time Frame: at 5 months
Population: Data was reported for month 5 from start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 129
units on a scale | 24.08 (17.23)

16. Secondary Outcome: Physical Health Quality of Life as Measured by a 12 Item Short-Form Health Survey
Description: Physical Health Quality of life measures were administered during screening and on Days 1 (±3), of Cycle 1, Day 1 (±3), of Cycle 2 and on day 1 (±7) of Cycles 3, 6, and then every 3 months thru Cycle 24 and at time of progression and /or end of treatment. SF-12 assesses aspects of quality of life including physical functioning, role functioning-physical, bodily pain, general health perceptions, vitality, social functioning, role functioning-emotional, and mental health. Subscale raw scores are transformed to put each subscale on a 0-100 range with higher scores indicative of greater functioning. Subscale scores are standardized based on US General Population norms and aggregated based on factor score coefficients into two component scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Component scores are norm-based t-scores meaning scores above 50 indicate better functioning than average functioning while scores below 50 indicate worse functioning.
Time Frame: up to 5 months
Population: Data was reported for month 5 from start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 126
units on a scale | 44.23 (11.31)

ADVERSE EVENTS:
Groups:
- Treatment (Ibrutinib): Patients treated with PCI-32765 capsules administered orally once daily at a dose of 420 mg for 28 day cycles. Weekly monitoring during the first month will occur followed by monthly evaluations for 2 additional months. Monitoring for patients at this point would be every 3 months with monthly CBC(complete blood count)and phone follow-up with a co-investigator on the study. A standard questionnaire will be used in this monthly phone assessment. Patients will continue to receive the study drug indefinitely as long as they are deriving clinical benefit (Complete Response or Partial Response or Stable Disease) and not experiencing any unacceptable toxicity. Subjects with disease progression will be removed from the study. Correlative laboratory samples, quality of life assessment, and immunologic data would be collected over time of therapy.
  ibrutinib: Patients received ibrutinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progres
Arm/Group | Treatment (Ibrutinib)
Serious Adverse Events (participants affected / at risk) | 152/152
Other Adverse Events (participants affected / at risk) | 152/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ibrutinib) (N=152)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Hemolytic Uremic Syndrome (Blood and lymphatic system disorders) | 1 (1)
Lymph Node Pain (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Cardiac Disorders-other (Cardiac disorders) | 1 (4)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Ventricular Arrythmia (Cardiac disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Colonic Perforation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Esophageal Ulcer (Gastrointestinal disorders) | 1 (1)
Gastric Hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Disorders-other (Gastrointestinal disorders) | 3 (4)
Jejunal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 (2)
Chills (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 5 (5)
Edema Limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 4 (4)
General Disorders and Administration Site Conditions - Other (General disorders) | 3 (3)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Sudden Death NOS (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (4)
Immune System Disorders - Other (Immune system disorders) | 1 (1)
Bone Infection (Infections and infestations) | 3 (3)
Bronchial Infection (Infections and infestations) | 4 (4)
Catheter Related Infection (Infections and infestations) | 2 (2)
Enterocolitis Infectious (Infections and infestations) | 3 (3)
Infections and Infestations-other (Infections and infestations) | 13 (16)
Lung Infection (Infections and infestations) | 32 (53)
Otitis Media (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 6 (7)
Sinusitis (Infections and infestations) | 1 (1)
Skin Infection (Infections and infestations) | 4 (4)
Soft Tissue Infection (Infections and infestations) | 2 (3)
Upper Respiratory Infection (Infections and infestations) | 5 (5)
Urinary Tract Infection (Infections and infestations) | 3 (8)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Injury, Poisoning and Procedural Complications - Other (Injury, poisoning and procedural complications) | 3 (3)
Intestinal Stoma Obstruction (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and Nutrition Disorders - Other (Metabolism and nutrition disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Weakness Left Sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and Connective Tissue Disorder - Other (Musculoskeletal and connective tissue disorders) | 3 (3)
Intracranial Hemorrhage (Nervous system disorders) | 2 (2)
Leukoencephalopathy (Nervous system disorders) | 2 (2)
Memory Impairement (Nervous system disorders) | 1 (1)
Nervous System Disorders - Other (Nervous system disorders) | 3 (4)
Syncope (Nervous system disorders) | 2 (2)
Transient Ischemic Attacks (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Psychiatric Disorders-Other (Psychiatric disorders) | 1 (1)
Renal and Urinary Disorders - Other (Renal and urinary disorders) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1)
Reproductive System and Breast Disorders - Other (Reproductive system and breast disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, Thoracic, and Mediastinal Disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and Medical Procedures - Other (Surgical and medical procedures) | 4 (4)
Hematoma (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Superior Vena Cava Syndrom (Vascular disorders) | 1 (1)
Thromboembolic Events (Vascular disorders) | 2 (2)
Vascular Disorders- Other (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ibrutinib) (N=152)
Anemia (Blood and lymphatic system disorders) | 43 (51)
Leukocytosis (Blood and lymphatic system disorders) | 25 (29)
Lymph node pain (Blood and lymphatic system disorders) | 14 (16)
Atrial Fibrillation (Cardiac disorders) | 13 (15)
Palpitations (Cardiac disorders) | 12 (15)
Sinus Bradycardia (Cardiac disorders) | 24 (28)
Sinus Tachycardia (Cardiac disorders) | 9 (11)
Ear and Labyrinth disorders (Ear and labyrinth disorders) | 10 (12)
Hearing impaired (Ear and labyrinth disorders) | 8 (8)
Vertigo (Ear and labyrinth disorders) | 8 (8)
Blurred vision (Eye disorders) | 19 (21)
Cataract (Eye disorders) | 13 (13)
Conjunctivitis (Eye disorders) | 8 (9)
Dry eye (Eye disorders) | 12 (13)
Eye Disorders (Eye disorders) | 35 (41)
Watering eyes (Eye disorders) | 8 (8)
Abdominal Pain (Gastrointestinal disorders) | 34 (39)
Bloating (Gastrointestinal disorders) | 24 (24)
Constipation (Gastrointestinal disorders) | 51 (66)
Diarrhea (Gastrointestinal disorders) | 100 (190)
Dry mouth (Gastrointestinal disorders) | 15 (15)
Dyspepsia (Gastrointestinal disorders) | 15 (17)
Dysphagia (Gastrointestinal disorders) | 10 (10)
Flatulence (Gastrointestinal disorders) | 17 (18)
Gastrointestional Disorder (Gastrointestinal disorders) | 73 (103)
Mucositis (Gastrointestinal disorders) | 70 (127)
Nausea (Gastrointestinal disorders) | 56 (86)
Oral Hemorrhage (Gastrointestinal disorders) | 28 (37)
Oral Pain (Gastrointestinal disorders) | 7 (8)
Stomach Pain (Gastrointestinal disorders) | 10 (10)
Vomiting (Gastrointestinal disorders) | 41 (59)
Chills (General disorders) | 36 (42)
Edema Limbs (General disorders) | 49 (59)
Fatigue (General disorders) | 83 (99)
Fever (General disorders) | 41 (55)
Flu Like Symptoms (General disorders) | 13 (15)
General Disorders (General disorders) | 27 (34)
Non-Cardiac chest pain (General disorders) | 12 (12)
Pain (General disorders) | 33 (42)
Bronchial Infection (Infections and infestations) | 18 (21)
Eye Infection (Infections and infestations) | 8 (9)
Infections and Infestations (Infections and infestations) | 32 (41)
Lung Infection (Infections and infestations) | 30 (43)
Nail Infection (Infections and infestations) | 9 (9)
Paronychia (Infections and infestations) | 11 (18)
Sinusitis (Infections and infestations) | 49 (68)
Skin Infection (Infections and infestations) | 35 (43)
Upper Respiratory Infection (Infections and infestations) | 72 (129)
Urinary Tract Infection (Infections and infestations) | 30 (52)
Bruising (Injury, poisoning and procedural complications) | 70 (93)
Fall (Injury, poisoning and procedural complications) | 20 (32)
Injury, Poisoning and procedural complications (Injury, poisoning and procedural complications) | 7 (7) — other
Lymphocyte count decreased (Investigations) | 25 (36)
Lymphocyte count increased (Investigations) | 70 (87)
Neutrophil count decreased (Investigations) | 80 (166)
Platelet count decreased (Investigations) | 44 (52)
Weight gain (Investigations) | 65 (75)
Weight loss (Investigations) | 39 (53)
White Blood cell decreased (Investigations) | 27 (38)
Anorexia (Metabolism and nutrition disorders) | 39 (39)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (30)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (9)
Hyperuricemia (Metabolism and nutrition disorders) | 17 (25)
Hypokalemia (Metabolism and nutrition disorders) | 9 (14)
Hyponatremia (Metabolism and nutrition disorders) | 14 (15)
Hypophosphatemia (Metabolism and nutrition disorders) | 12 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 56 (77)
Arthritis (Musculoskeletal and connective tissue disorders) | 24 (26)
Back pain (Musculoskeletal and connective tissue disorders) | 37 (41)
Bone pain (Musculoskeletal and connective tissue disorders) | 12 (12)
Musculoskeletal and Connective tissue disorder-other (Musculoskeletal and connective tissue disorders) | 104 (123)
Myalgia (Musculoskeletal and connective tissue disorders) | 29 (34)
Neck pain (Musculoskeletal and connective tissue disorders) | 9 (10)
Pain Extremity (Musculoskeletal and connective tissue disorders) | 29 (34)
Neoplasms benign, malignant and unspecified-other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 37 (49)
Dizziness (Nervous system disorders) | 55 (69)
Dysgeusia (Nervous system disorders) | 17 (18)
Headache (Nervous system disorders) | 63 (79)
Nervous System Disorders-other (Nervous system disorders) | 10 (10)
Paresthesia (Nervous system disorders) | 48 (54)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Informed Consent Form (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT01589302/ICF_000.pdf